CLINICAL TRIAL: NCT04043923
Title: A Phase 2b Double-blind, Randomized, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of Norketotifen (NKT) in the Treatment of Acute Uncomplicated Influenza-like Illness (ILI)
Brief Title: Norketotifen for the Treatment of Uncomplicated Influenza-like Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKT-202
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Influenza -Like Illness
MeSH Terms: interventions — norketotifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Norketotifen (Experimental): Norketotifen oral capsules, once daily for 5 days
  Interventions: Drug: Norketotifen
- Placebo (Placebo Comparator): Placebo oral capsules, once daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norketotifen — Oral capsule
  Arms: Norketotifen
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2b, multi-center, double-blind, randomized, placebo-controlled, parallel-group study of NKT versus placebo in otherwise healthy adults presenting with acute uncomplicated ILI due to influenza or other respiratory viruses in a community setting.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and comply with all study procedures, and willing to provide written informed consent prior to the pre-dose examinations
2. Symptoms of ILI including all of the following:

   * Fever ≥38º Celsius (oral) in the predose examinations or >4 hours after dosing of antipyretics if they were taken
   * At least one of the following general systemic symptoms associated with ILI are present with a severity of moderate or greater: headache, feverishness or chills, muscle or joint pain, fatigue
   * At least one of the following respiratory symptoms associated with ILI are present with a severity of moderate or greater: cough, sore throat, nasal congestion
3. The time interval between the onset of symptoms and the predose examinations is ≤96 hours. The onset of symptoms is defined as either:

   * Time of the first increase in body temperature (an increase of at least 1º Celsius from normal body temperature)
   * Time when the subject experiences at least one general or respiratory symptom
4. Females of childbearing potential and males agree to use an appropriate method of contraception as detailed in the protocol

Exclusion Criteria:

1. Female subjects who are pregnant, 2 weeks post-partum, or breastfeeding
2. Severe ILI requiring inpatient treatment
3. Any of the following risk factors (according to the CDC's list of People at High Risk for Developing Serious Flu-Related Complications):

   * Residents of nursing homes or other long-term care facilities
   * American Indians and Alaska natives
   * Asthma
   * Chronic lung disease (such as chronic obstructive pulmonary disease or cystic fibrosis)
   * Neurological and neurodevelopmental conditions (including disorders of the brain, spinal cord, peripheral nerve, and muscle such as cerebral palsy, epilepsy [seizure disorders], stroke, intellectual disability, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury)
   * Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease)
   * Blood disorders (such as sickle cell disease)
   * Endocrine disorders (such as diabetes mellitus)
   * Kidney disorders
   * Liver disorders
   * Metabolic disorders (such as inherited metabolic disorders and mitochondrial disorders)
   * Compromised immune system due to disease or medication (such as subjects with human immunodeficiency virus or cancer, or those on chronic steroids)
   * Extreme obesity (body mass index ≥40 kg/m^2)
4. Presence of any severe or uncontrolled medical or psychiatric illness
5. History of or current autoimmune disease
6. History of recurrent lower respiratory tract infection
7. Any concurrent infection requiring systemic antimicrobial and/or antiviral therapy
8. Female subjects who are pregnant or breastfeeding
9. Any clinically significant electrocardiogram test
10. Received baloxavir, oseltamivir, peramivir, zanamivir, rimantadine, or amantadine within 30 days prior to the pre-dose examinations
11. Received an investigational monoclonal antibody for a viral disease in the last year prior to the pre-dose examinations
12. Received ketotifen fumarate, cromolyn sodium, or nedocromil sodium by any route of administration within 30 days prior to the pre-dose examinations
13. Exposure to an investigational drug within 30 days prior to the pre-dose examinations
14. History of allergic reaction to ketotifen
15. Any prior exposure to norketotifen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of symptoms | 14 days
  Time to alleviation of the symptoms of ILI (headache, feverishness/chills, muscle/joint pain, fatigue, cough, sore throat, nasal congestion)

SECONDARY OUTCOMES:
Proportion of subjects whose symptoms have been alleviated at each time point through Day 5 | 5 days
Change from baseline in composite symptom score at each time point through Day 5 | 5 days
Time to resolution of fever (body temperature equal to or less than 37ºC) | 14 days
Body temperature at each time point through Day 5 | 5 days
Time to alleviation of individual symptoms (headache, feverishness/chills, muscle/joint pain, fatigue, cough, sore throat, nasal congestion) | 14 days
Time to resumption of normal activity | 14 days
Use of rescue medication (acetaminophen) | 14 days

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Cahaba Research, Birmingham, Alabama
  - Precision Trials AZ, Phoenix, Arizona
  - Long Beach Clinical Trial Services, Long Beach, California
  - Empire Clinical Research, Pomona, California
  - Northern California Research, Sacramento, California
  - AFC Urgent Care, Denver, Colorado
  - South Florida Research Center, Miami, Florida
  - Premier Research Associate, Miami, Florida
  - Gulfcoast Medical Research, Tampa, Florida
  - DelRicht Research, Baton Rouge, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - The Clinical Research Center, St Louis, Missouri
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Health Concepts, Rapid City, South Dakota
  - Premier Family Physicians, Austin, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - CityDoc Urgent Care, Dallas, Texas
  - Village Health Partners, Plano, Texas

IPD SHARING:
Plan to Share IPD: No